CLINICAL TRIAL: NCT03155516
Title: Evaluation of the Effect of Good Pain Management (GPM) Ward Program on Pattern of Care and Patient-Reported Outcomes of Moderate to Severe Cancer Pain Patients
Brief Title: Effect of Good Pain Management (GPM) Ward Program on Moderate to Severe Cancer Pain Patients
Acronym: GPM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taiwan Mundipharma Pharmaceuticals Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: GPM16-TW-401
Record Dates: First submitted 2017-05-14; First posted 2017-05-16 (Actual); Last update posted 2017-05-16 (Actual); Status verified 2017-05

CONDITIONS: Cancer; Pain
Keywords: Cancer pain; GPM; pain assessment
MeSH Terms: conditions — Neoplasms; Pain; Cancer Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GPM Ward (Experimental): Good Pain management ward
  Interventions: Other: Good pain management (GPM) procedure
- Control Ward (Active Comparator): Current practice controlled ward
  Interventions: Other: Current practice procedure

INTERVENTIONS:
Other: Good pain management (GPM) procedure — In the GPM ward, a close pain assessment will be carried within 1 hour after admission. After the assessment, patient will be given analgesic treatment as needed, by acceptable route, frequency and dosage. A good titration is required in GPM ward. Patient will be close monitor his/her pain level regarding pain score. In opioid use, when patient complains patient level ≥ 4, low dose strong opioids will be introduced in patient suffering with moderate pain.
  Compare with current practice, GPM ward will perform pain assessment with higher frequency for adjusting of analgesic medications if required.
  Arms: GPM Ward
Other: Current practice procedure — Current practice clinical procedure for pain management
  Arms: Control Ward

SUMMARY:
This study aims to set up a standardized cancer pain ward - known as the Good Pain Management (GPM) Ward with streamlined assessment and management procedures to act as a pain management model. In particular, it will enforce regular pain assessment from and throughout hospital admission, and treatment protocols introducing the use of strong-opioids in moderate cancer pain patients, following National Cancer Care Network (NCCN) Adult Cancer Pain Guidelines. The GPM ward will be compared against current-practice controlled ward.

DETAILED DESCRIPTION:
This is a double-arm, randomized, multi-center, current practice-controlled study. Approximately 150 cancer pain patients with collecting questionnaires admitted to an inpatient department from 3 national hospitals: Kaohsiung Medical University Hospital, Kaohsiung Municipal Ta-Tung Hospital and Kaohsiung Municipal HsiaoKang Hospital will be invited into this study. Eligible patients will be randomized to one of the following pain control wards in a 1:1 ratio.

* GPM Ward: Good Pain management ward
* Control Ward: Current practice-controlled ward Surveys, pain level measurements and dosage used will be collected in 48±8 hours. The pain management index (PMI) will be assessed as primary objective. The patient satisfaction, outcome questionnaire (APS-POQ) and SF-36 will be assessed in secondary objectives.

Once patient is admitted to the ward and agrees to participate in the study, the patient will be randomly and blindly assigned to either GPM ward or Control Ward. In the Control Ward, patient will receive the current practice of pain management, with less assessment procedure.

This study will investigate the benefits and effect of good pain control on patient outcomes in hospitalized cancer pain patients. The results aim to demonstrate the viability of GPM ward in daily practices and its measurable impact on the patient outcomes including patient treatment satisfaction as well as quality of life.

1. Primary objectives:

   • To assess pain management index (PMI)
2. Secondary objectives:

(1) To assess the satisfaction of pain control during admission (2) To analyze the Patient Outcome Questionnaire (APS-POQ) (3) To analyze the SF-36 Questionnaire

ELIGIBILITY:
Inclusion Criteria:

1. Females and males aged ≥ 20
2. Understand Chinese/Taiwanese and able to finish the questionnaire
3. Alert enough to respond and understand
4. Hospitalized for ≥ 24 hours
5. ECOG ≤ 2
6. Cancer patients with cancer-related pain

Exclusion Criteria:

1. Patient diagnosed with non-cancer pain or unexplained pain
2. Patient with moderate to severe mental disorder
3. Patient receiving operation or invasive procedure within 24 hours before admission

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2016-08-30 (Actual); Primary Completion 2019-08-29 (Estimated); Study Completion 2019-08-29 (Estimated)

PRIMARY OUTCOMES:
Pain management index (PMI) assessment | Up to 56 hours
  The change of mean PMI score, pain-reporting rate and adequacy of pain treatment using pain management index

SECONDARY OUTCOMES:
Satisfaction of pain control during admission | Up to 56 hours
  Patient satisfaction about pain control
Patient outcome questionnaire (APS-POQ) analysis | Up to 56 hours
  The analysis of APS-POQ outcome
SF-36 Questionnaire analysis | Up to 24 hours in screening period
  The analysis of SF-36

CONTACTS AND LOCATIONS:
Overall Officials: Jaw-Yuan Wang, PhD, Principal Investigator — Kaohsiung Medical University Chung-Ho Memorial Hospital
Locations (3):
- Taiwan (3):
  - Kaohsiung Municipal Ta-Tung Hospital, Kaohsiung City
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Kaohsiung Municipal Siaogang Hospital, Kaohsiung City

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kurita GP, Tange UB, Farholt H, Sonne NM, Stromgren AS, Ankersen L, Kristensen L, Bendixen L, Gronvold M, Petersen MA, Nordly M, Christrup L, Niemann C, Sjogren P. Pain characteristics and management of inpatients admitted to a comprehensive cancer centre: a cross-sectional study. Acta Anaesthesiol Scand. 2013 Apr;57(4):518-25. doi: 10.1111/aas.12068. Epub 2013 Jan 22. PMID 23336265
- [Background] Sharma N, Hansen CH, O'Connor M, Thekkumpurath P, Walker J, Kleiboer A, Murray G, Espie C, Storey D, Sharpe M, Fleming L. Sleep problems in cancer patients: prevalence and association with distress and pain. Psychooncology. 2012 Sep;21(9):1003-9. doi: 10.1002/pon.2004. Epub 2011 Jul 1. PMID 21726015
- [Background] American Society of Anesthesiologists Task Force on Chronic Pain Management; American Society of Regional Anesthesia and Pain Medicine. Practice guidelines for chronic pain management: an updated report by the American Society of Anesthesiologists Task Force on Chronic Pain Management and the American Society of Regional Anesthesia and Pain Medicine. Anesthesiology. 2010 Apr;112(4):810-33. doi: 10.1097/ALN.0b013e3181c43103. No abstract available. PMID 20124882
- [Background] Ripamonti CI, Bandieri E, Roila F; ESMO Guidelines Working Group. Management of cancer pain: ESMO Clinical Practice Guidelines. Ann Oncol. 2011 Sep;22 Suppl 6:vi69-77. doi: 10.1093/annonc/mdr390. No abstract available. PMID 21908508
- [Background] National Comprehensive Cancer Network. Adult cacner pain
- [Background] Tang ST, Tang WR, Liu TW, Lin CP, Chen JS. What really matters in pain management for terminally ill cancer patients in Taiwan. J Palliat Care. 2010 Autumn;26(3):151-8. PMID 21047037
- [Background] Liang SY, Li CC, Wu SF, Wang TJ, Tsay SL. The prevalence and impact of pain among Taiwanese oncology outpatients. Pain Manag Nurs. 2011 Dec;12(4):197-205. doi: 10.1016/j.pmn.2010.10.034. Epub 2011 Jan 28. PMID 22117751
- [Background] Seya MJ, Gelders SF, Achara OU, Milani B, Scholten WK. A first comparison between the consumption of and the need for opioid analgesics at country, regional, and global levels. J Pain Palliat Care Pharmacother. 2011;25(1):6-18. doi: 10.3109/15360288.2010.536307. PMID 21426212
- [Background] Duthey B, Scholten W. Adequacy of opioid analgesic consumption at country, global, and regional levels in 2010, its relationship with development level, and changes compared with 2006. J Pain Symptom Manage. 2014 Feb;47(2):283-97. doi: 10.1016/j.jpainsymman.2013.03.015. Epub 2013 Jul 17. PMID 23870413
- [Background] Pan HH, Ho ST, Lu CC, Wang JO, Lin TC, Wang KY. Trends in the consumption of opioid analgesics in Taiwan from 2002 to 2007: a population-based study. J Pain Symptom Manage. 2013 Feb;45(2):272-8. doi: 10.1016/j.jpainsymman.2012.02.014. Epub 2012 Aug 11. PMID 22889859
- [Background] Wang CH, Lee SY. Undertreatment of caner pain. Acta Anaesthesiol Taiwan. 2015 Jun;53(2):58-61. doi: 10.1016/j.aat.2015.05.005. Epub 2015 Jun 7. PMID 26063333
- [Derived] Su WC, Chuang CH, Chen FM, Tsai HL, Huang CW, Chang TK, Hou MF, Wang JY. Effects of Good Pain Management (GPM) ward program on patterns of care and pain control in patients with cancer pain in Taiwan. Support Care Cancer. 2021 Apr;29(4):1903-1911. doi: 10.1007/s00520-020-05656-x. Epub 2020 Aug 15. PMID 32803728